CLINICAL TRIAL: NCT00584987
Title: A Combination of Intranasal Steroid/Oxymetazoline Leads to Faster Relief of Nasal Congestion Without Inducing Rhinitis Medicamentosa
Brief Title: Intranasal Steroids and Oxymetazoline in Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Robert Naclerio, MD, University of Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15059B
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Results first posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-10

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — fluticasone furoate; Fluticasone; Oxymetazoline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo FF + Placebo OXY (Placebo Comparator): Placebo Fluticasone furoate + Placebo Oxymetazoline, 2 puffs of each nasal spray in each nostril in the pm
  Interventions: Drug: Placebo Fluticasone furoate; Drug: Placebo Oxymetazoline
- FF + Placebo OXY (Active Comparator): Fluticasone furoate + Placebo Oxymetazoline, 2 puffs of each nasal spray in each nostril in the pm
  Interventions: Drug: Fluticasone furoate; Drug: Placebo Oxymetazoline
- Placebo FF + OXY (Active Comparator): Placebo Fluticasone furoate + Oxymetazoline, 2 puffs of each nasal spray in each nostril in the pm
  Interventions: Drug: Placebo Fluticasone furoate; Drug: Oxymetazoline
- FF + OXY (Active Comparator): Fluticasone furoate + Oxymetazoline, 2 puffs of each nasal spray in each nostril in the pm
  Interventions: Drug: Fluticasone furoate; Drug: Oxymetazoline

INTERVENTIONS:
Drug: Fluticasone furoate — 2 puffs of each nasal spray in each nostril in the pm
  Other Names: Veramyst
  Arms: FF + OXY; FF + Placebo OXY
Drug: Placebo Fluticasone furoate — 2 puffs of each nasal spray in each nostril in the pm
  Arms: Placebo FF + OXY; Placebo FF + Placebo OXY
Drug: Oxymetazoline — 2 puffs of each nasal spray in each nostril in the pm
  Other Names: Oxymetazoline hydrochloride
  Arms: FF + OXY; Placebo FF + OXY
Drug: Placebo Oxymetazoline — 2 puffs of each nasal spray in each nostril in the pm
  Arms: FF + Placebo OXY; Placebo FF + Placebo OXY

SUMMARY:
We hypothesize that once daily use of oxymetazoline will not cause significant rhinitis medicamentosa and that the combination of fluticasone furoate plus oxymetazoline leads to faster relief of nasal congestion secondary to perennial allergic rhinitis than the use of fluticasone furoate alone.

DETAILED DESCRIPTION:
We performed a 6-week, 4-group, parallel, randomized, double-blind, double-dummy, clinical trial in 60 patients with perennial allergic rhinitis. After an initial screening with an allergy questionnaire and skin puncture testing to confirm an allergic response to a perennial allergen (cat, dog, dust mite, indoor mold), qualified individuals were randomized into 1 of 4 treatment groups. The 4 groups received the following treatments: placebo, OXY (0.05%, 2 puffs in each nostril every evening), FF nasal spray (110 mg per day), and FF nasal spray plus OXY (FF/OXY). All participants received 2 nasal sprays at night, with 1 spray containing FF or its placebo, the other oxymetazoline or its placebo. The nasal sprays were labeled with participant code numbers, and the investigator assigned participants in a sequential randomized fashion to a study code number in blocks of 4. Dropouts were replaced until 60 subjects were randomized. Replacement subjects were assigned the next sequential treatment. Thus, the number of subjects in each group was not exactly 15.

Eligible participants completed the Rhinitis Quality of Life Questionnaire (RQLQ) and underwent measurement of nasal volume by acoustic rhinometry before starting the study. Participants were instructed to keep a diary of daily symptoms, nasal peak inspiratory flow (NPIF) meter readings, and medication use during the study; no rescue medications were allowed. The severity of sneezing, rhinorrhea, nasal congestion, and other symptoms was recorded in the morning (reflective of symptoms overnight) and evening (reflective of daytime symptoms) on a 0 to 3 scale. Intake of the study medication was performed once daily, at night, after recording of symptoms and NPIF values. Subjects returned to the nasal laboratory every 2 weeks for a total of 4 weeks for review of the symptom diaries, replacement of medications, performance of acoustic rhinometry, and completion of the RQLQ. After the fourth week, participants stopped treatment, returned medication, and continued with the clinical trial for 2 additional weeks. During this time, they maintained symptom diaries and NPIF measurements twice daily. At the end of the 2-week period, participants returned to the nasal laboratory to perform a final acoustic rhinometry, complete an RQLQ survey, and return the diaries.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 55 years of age.
2. History of perennial allergic rhinitis.
3. Positive skin test to dust mite, dog, cat or indoor mold antigen.
4. And a combined nasal morning and evening score of ≥4 for nasal congestion in the day preceding entry

Exclusion Criteria:

1. Physical signs or symptoms suggestive of renal, hepatic or cardiovascular disease.
2. Pregnant or lactating women.
3. Subjects treated with systemic steroids during the previous 30 days.
4. Subjects treated with topical (inhaled, intranasal or intraocular) steroids, Nasalcrom or Opticrom during the previous 30 days.
5. Subjects treated with oral antihistamine/decongestants during the previous seven days.
6. Subjects treated with topical (intranasal or intraocular) antihistamine/decongestants during the previous 3 days.
7. Subjects treated with immunotherapy and are escalating their dose.
8. Subjects on chronic anti-asthma medications.
9. Subjects with polyps in the nose or a significantly displaced septum.
10. Upper respiratory infection within 14 days of study start.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Baroody FM, Brown D, Gavanescu L, DeTineo M, Naclerio RM. Oxymetazoline adds to the effectiveness of fluticasone furoate in the treatment of perennial allergic rhinitis. J Allergy Clin Immunol. 2011 Apr;127(4):927-34. doi: 10.1016/j.jaci.2011.01.037. Epub 2011 Mar 5. PMID 21377716

RESULTS

PARTICIPANT FLOW:
Groups:
- PL FF + PL OXY: Placebo Fluticasone furoate + Placebo Oxymetazoline, 2 puffs of each nasal spray in each nostril in the pm
- FF + PL OXY: Fluticasone furoate + Placebo Oxymetazoline, 2 puffs of each nasal spray in each nostril in the pm
- PL FF + OXY: Placebo Fluticasone furoate + Oxymetazoline, 2 puffs of each nasal spray in each nostril in the pm
Period: Overall Study
Arm/Group | PL FF + PL OXY | FF + PL OXY | PL FF + OXY | FF + OXY
Started | 15 | 16 | 17 | 16
Completed | 14 | 15 | 16 | 15
Not Completed | 1 | 1 | 1 | 1
Not completed — Protocol Violation | 1 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo FF + Placebo OXY | FF + Placebo OXY | Placebo FF + OXY | FF + OXY | Total
Number analyzed (Participants) | 15 | 16 | 17 | 16 | 64
Age Continuous [Mean (Standard Deviation); unit: years] | 29.6 (11) | 31.7 (9.5) | 26.6 (5.2) | 28.6 (8.7) | 28.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 10 | 9 | 41
  Male | 5 | 4 | 7 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Total Nasal Congestion Symptom Score
Description: The severity of nasal congestion was recorded in the morning (reflective of symptoms overnight) and evening (reflective of daytime symptoms) on a 0 to 3 scale. The total nasal congestion symptom score was obtained by adding the symptoms obtained on all 28 days of treatment. Values for this outcome are in the range of 0 to 168 (i.e., 6 x 28). Congestion scores increase with congestion severity (i.e., higher numbers correspond to worse congestion).
Time Frame: 28 days of treatment
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo FF + Placebo OXY | FF + Placebo OXY | Placebo FF + OXY | FF + OXY
Number analyzed (Participants) | 14 | 15 | 16 | 15
units on a scale | 94 [60 to 157] | 70 [34 to 151] | 75 [7 to 132] | 68 [2 to 115]

2. Secondary Outcome: RQLQ Score [Baseline]
Description: The Rhinoconjunctivitis Quality-of-Life Questionnaire (RQLQ) has 28 questions and focusses on 7 domains that may be significantly impaired in participants with seasonal allergic rhinoconjunctivitis: sleep impairment, non-nasal symptoms, practical problems, nasal symptoms, eye symptoms, activity limitations, and emotional difficulty. The RQLQ score is the mean of all 28 responses and the individual domain scores are the means of the items in those domains. RQLQ scores range from 0-6, with a higher score indicating more significant impairment.
Time Frame: assessed at baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo FF + Placebo OXY | FF + Placebo OXY | Placebo FF + OXY | FF + OXY
Number analyzed (Participants) | 14 | 15 | 16 | 15
units on a scale | 3.07 (0.28) | 3.25 (0.29) | 2.99 (0.28) | 2.60 (0.22)

3. Secondary Outcome: RQLQ Score [2 Weeks]
Description: as for outcome 2
Time Frame: assessed 2 weeks after initiation of treatment regimen
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo FF + Placebo OXY | FF + Placebo OXY | Placebo FF + OXY | FF + OXY
Number analyzed (Participants) | 14 | 15 | 16 | 15
units on a scale | 2.20 (0.26) | 2.03 (0.26) | 2.11 (0.20) | 1.62 (0.24)

4. Secondary Outcome: RQLQ Score [4 Weeks]
Description: as for outcome 2
Time Frame: assessed 4 weeks after initiation of treatment regimen
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo FF + Placebo OXY | FF + Placebo OXY | Placebo FF + OXY | FF + OXY
Number analyzed (Participants) | 14 | 15 | 16 | 15
units on a scale | 1.75 (0.24) | 1.37 (0.24) | 1.85 (0.20) | 1.26 (0.22)

5. Secondary Outcome: RQLQ Score [6 Weeks]
Description: as for outcome 2
Time Frame: assessed 6 weeks after initiation of treatment regimen
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo FF + Placebo OXY | FF + Placebo OXY | Placebo FF + OXY | FF + OXY
Number analyzed (Participants) | 14 | 15 | 16 | 15
units on a scale | 1.85 (0.25) | 1.83 (0.33) | 2.03 (0.27) | 1.55 (0.19)

6. Secondary Outcome: Total NPIF
Description: Nasal peak inspiratory flow (NPIF) is a physiological measure of nasal airflow which is particularly sensitive to nasal valve collapse. NPIF was measured objectively in liters per minute with an In-Check Peak Inspiratory FlowMeter (Ferraris Medical Inc, Orchard Park, NY). Subjects obtained 3 readings every morning and every evening and recorded the best flow measured. The morning and evening NPIF measurements were summed for days 2 through 28 of the treatment cycle, yielding the total NPIF outcome measure. NPIF scores increase with air flow quality (i.e., higher NPIF values are indicative of better nasal air flow).
Time Frame: days 2 through 28 of the treatment cycle
Measure: Median (Full Range); unit: liters per minute
Arm/Group | Placebo FF + Placebo OXY | FF + Placebo OXY | Placebo FF + OXY | FF + OXY
Number analyzed (Participants) | 14 | 15 | 16 | 15
liters per minute | 5240 [2370 to 9085] | 5680 [3890 to 9715] | 4485.5 [3270 to 7840] | 5520 [3322 to 10280]

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events 2 weeks after treatment as outlined in the protocol. No subjects presented with adverse events after the official follow-up period concluded.
Arm/Group | Placebo FF + Placebo OXY | FF + Placebo OXY | Placebo FF + OXY | FF + OXY
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 2/15 | 4/16 | 2/17 | 2/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo FF + Placebo OXY (N=15) | FF + Placebo OXY (N=16) | Placebo FF + OXY (N=17) | FF + OXY (N=16)
Headaches (General disorders) | 2 | 4 | 2 | 2 — A headache or cephalalgia is pain anywhere in the region of the head or neck.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes